CLINICAL TRIAL: NCT00804895
Title: A Double Blind Randomized Controlled Trial of Greater Occipital Nerve Infiltration in Cluster Headache
Brief Title: Cluster Headache Cortivazol Injection (CHCI)
Acronym: CHCI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P080602
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Cluster Headache
Keywords: cluster headache; greater occipital nerve block; cortivazol
MeSH Terms: conditions — Cluster Headache | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): subcutaneous injection of Cortivazol ALTIM, 3,375mg
  Interventions: Drug: ALTIM, cortivazol injections; Drug: Verapamil
- 2 (Placebo Comparator): PROAMP, subcutaneous serum physiological saline
  Interventions: Drug: PROAMP, subcutaneous serum physiological saline; Drug: Verapamil

INTERVENTIONS:
Drug: ALTIM, cortivazol injections — ALTIM, cortivazol in greater occipital nerve injection separated by 2 or 3 days each.
  Other Names: ALTIM, cortivazol injections greater occipital
  Arms: 1
Drug: PROAMP, subcutaneous serum physiological saline — Three injections will be performed at the level of the greater occipital nerve with a suboccipital approach. Injection will be separated by two or three days each.
  Arms: 2
Drug: Verapamil — standard prophylactic treatment

SUMMARY:
the aim of tis study is to demonstrate the efficacy of cortivazol injections at the level of the greater occipital nerve to diminish the frequency of cluster headache (episodic or chronic) attacks during an active period. Injections will be used in adjunct with oral verapamil.

DETAILED DESCRIPTION:
Cluster headache is characterized by unilateral attacks of severe periorbital pain accompanied by autonomic symptoms and restlessness. Though patients may respond to the standard prophylactic treatment of verapamil, some are refractory and continue to suffer from numerous attacks, with a limit of two doses of subcutaneous sumatriptan per day. Some patients also have contra-indications to standard prophylactic or acute treatments. Other preventive treatments like systemic steroids, lithium and methysergide may cause significant side effects. We intend to show the efficacy of occipital nerve injections with cortivazol, in adjunct to verapamil, in cluster headache patients. We expect a diminution of attack frequency over two weeks, with a protocol of three injections separated by two or three days each. Tolerance and safety will be examined.

ELIGIBILITY:
Inclusion Criteria:

* patient age, man or woman whose age is between 18 and 65 included
* patient who signed a free express and informed consent
* patient with cluster headache, episodic or chronic according to the criteria of International Headache Society (ICHD-II)
* patient with more than two episodes of CH per day
* patient with a normal medical examination

Exclusion Criteria:

* patient not affiliated with a social security scheme (or beneficiary entitled)
* patient with another diagnosis ICHD-II,and being unable to differentiate CH attacks from its other cranial pain
* patient of CH having started his episodic active period more than 30 days ago
* patient with a contra-indication to verapamil
* patient with a known allergy to cortivazol
* patient with anticoagulant therapy or having a bleeding disorder
* patient unable to complete the schedule crisis
* patient non-compliant or unable to follow the research protocol
* women without contraception, pregnant, or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with a daily attack frequency equal or inferior to two for the period going from two days after third injection to four days after the third injection | 2009

SECONDARY OUTCOMES:
total number of attacks on the J1-J15 period | 2009
percentage of patients with a 50% or more decrease in attacks frequency at J15 | 2009
percentage of patients reaching a remission at J30 defined as an absence of attacks for seven days or more | 2009
interval between the first injection and appearance of a remission | 2009
percentage of patients suffering from chronic CH, having reached a daily attack frequency equal or inferior to two, presenting a recurrence of attacks after J15, defined as more than two attacks per day | 2009
number of patients (episodic or chronic) presenting a daily attack frequency equal or inferior to two at J30 | 2009
number of chronic patients presenting a daily attack frequency equal or inferior to two at J90 | 2009
HIT-6 scores, comparison between groups at J0 and J30 | 2009
tolerance of treatment : percentage of patients showing side effects | 2009
safety of treatment: percentage of patients with serious adverse events | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Dominique VALADE, MD, Principal Investigator — CHU Lariboisière, AP-HP
Locations (1):
- CHU Lariboisière, AP-HP, Centre des Urgences Céphalées (Emergency Headacha Center), Paris, Île-de-France Region, France

REFERENCES:
- [Result] Leroux E, Valade D, Taifas I, Vicaut E, Chagnon M, Roos C, Ducros A. Suboccipital steroid injections for transitional treatment of patients with more than two cluster headache attacks per day: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2011 Oct;10(10):891-7. doi: 10.1016/S1474-4422(11)70186-7. Epub 2011 Sep 6. PMID 21903477